CLINICAL TRIAL: NCT01666808
Title: Advanced Molecular Imaging With Anti-3-[18F]FACBC PET-CT to Improve the Selection and Outcomes of Prostate Cancer Patients Receiving Post-prostatectomy Radiotherapy
Brief Title: FACBC Outcomes for Post Prostatectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ashesh B Jani, Professor & Residency Program Director, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057680; 1R01CA169188-01 (NIH)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FACBC PET scan (Experimental): A trial group in which anti-3-[18F]FACBC PET-CT is used to guide radiotherapy decisions and radiotherapy treatment volumes.
  Interventions: Drug: FACBC
- Conventional-Only Imaging (Active Comparator): A control group whose treatment decisions will be made based on conventional imaging - bone scan and abdominopelvic CT and/or MR scan.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Drug: FACBC — FACBC is given intravenously prior to PET scan, radiotherapy decisions and treatment guided by PET findings
  Other Names: anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid
  Arms: FACBC PET scan
Radiation: Radiation therapy — External beam radiotherapy to prostate bed +/- pelvic lymph nodes; final dose of 66.6 Gy.
  Other Names: Intensity-modulated radiotherapy (IMRT)
  Arms: Conventional-Only Imaging

SUMMARY:
Investigators will perform a study with 162 patients in whom there is a strong suspicion of prostate cancer that has returned to the body after having a prostatectomy. Half of these patients will have radiotherapy decision-making and delivery per the usual routine, and half of these patients will have the radiotherapy decision and volumes guided by the FACBC test (anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (anti-3- [18F]FACBC). The major goal of the investigation is to see whether the FACBC improves the selection and the cancer control rates of post-surgery patients with a rising PSA who undergo radiotherapy.

DETAILED DESCRIPTION:
Prostate cancer is the most common solid tumor, with approximately 200,000 new cases diagnosed per year. Several different local therapies are available for treatment, including surgery and radiotherapy Significant advances have been made in the technical aspects of surgery and of radiotherapy which have improved both the cancer control outcomes as well as the morbidity of treatment. Despite these significant advances, approximately 30% of patients treated with definitive local therapy experience recurrent disease. Recurrent disease after prostatectomy usually manifests with rising PSA (blood test for prostate cancer). The PSA level is often of limited use in differentiating local recurrence (ie. recurrence in the prostate bed) from recurrence outside of the prostate bed ( extra-prostatic recurrence).

One PET radiotracer which has shown promise in the staging and restaging of patients with prostate carcinoma is anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (anti-3-[18F]FACBC) which is a synthetic amino acid analog. FACBC demonstrated higher accuracy compared with 111Indium-capromab-pendetide in the restaging of patients with suspected recurrent prostate carcinoma.

The major goal in this proposed investigation is to use advanced molecular imaging to better guide post-prostatectomy decision making, in terms of guiding the decision to deliver radiotherapy, and in terms of the exact areas treated with radiotherapy.

Investigators will perform a study with 162 patients in whom there is a strong suspicion of prostate cancer that has returned to the body after having a prostatectomy. Half of these patients will have radiotherapy decision-making and delivery per the usual routine, and half of these patients will have the radiotherapy decision and volumes guided by the FACBC test. The major goal of the investigation is to see whether the FACBC improves the selection and the cancer control rates of post-surgery patients with a rising PSA who undergo radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, post radical-prostatectomy Detectable PSA
* ECOG/Zubrod Performance Status of 0-2
* Negative technetium 99-m MDP or F-18 PET bone scan for skeletal metastasis
* CT or MR scan of abdomen and pelvis which does not suggest presence of metastatic disease outside of the pelvis
* Willingness to undergo pelvic radiotherapy.

Exclusion Criteria:

* Contraindications to radiotherapy (including active inflammatory bowel disease or prior pelvic XRT)
* Inability to undergo anti-3-[18F]FACBC PET-CT
* Age under 18
* Metastatic disease outside of pelvis on any imaging or biopsy
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Severe acute co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization in the last 3 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh B Jani, MD, MSEE, Principal Investigator — Emory University; David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jani AB, Schreibmann E, Goyal S, Halkar R, Hershatter B, Rossi PJ, Shelton JW, Patel PR, Xu KM, Goodman M, Master VA, Joshi SS, Kucuk O, Carthon BC, Bilen MA, Abiodun-Ojo OA, Akintayo AA, Dhere VR, Schuster DM. 18F-fluciclovine-PET/CT imaging versus conventional imaging alone to guide postprostatectomy salvage radiotherapy for prostate cancer (EMPIRE-1): a single centre, open-label, phase 2/3 randomised controlled trial. Lancet. 2021 May 22;397(10288):1895-1904. doi: 10.1016/S0140-6736(21)00581-X. Epub 2021 May 7. PMID 33971152
- [Result] Dhere VR, Schuster DM, Goyal S, Schreibmann E, Hershatter BW, Rossi PJ, Shelton JW, Patel PR, Jani AB. Randomized Trial of Conventional Versus Conventional Plus Fluciclovine (18F) Positron Emission Tomography/Computed Tomography-Guided Postprostatectomy Radiation Therapy for Prostate Cancer: Volumetric and Patient-Reported Analyses of Toxic Effects. Int J Radiat Oncol Biol Phys. 2022 Aug 1;113(5):1003-1014. doi: 10.1016/j.ijrobp.2022.04.005. Epub 2022 Apr 11. PMID 35417762

RESULTS

PARTICIPANT FLOW:
Groups:
- FACBC PET Scan: A trial group in which anti-3-[18F]FACBC PET-CT is used to guide radiotherapy decisions and radiotherapy treatment volumes.
  FACBC: FACBC is given intravenously prior to PET scan
Period: Overall Study
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Started | 83 | 82
Completed | 67 | 66
Not Completed | 16 | 16
Not completed — Lost to Follow-up | 9 | 15
Not completed — Withdrawal by Subject | 3 | 1
Not completed — No radiotherapy given, due to extrapelvic uptake on PET scan | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FACBC PET Scan | Conventional-Only Imaging | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Median (Full Range); unit: years] | 61 [42 to 75] | 61 [46 to 78] | 61 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 83 | 82 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 29 | 59
  White | 52 | 52 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 82 | 165
Gleason score ≥8 [Count of Participants; unit: Participants] — Pathological grade was measured on the prostatectomy specimen. Gleason Grading goes from 2 thru 10, with higher scores being worse prognostically. Gleason scores of 8 and higher are considered high-grade, so this measure was designed to see whether the percentage of high-grade patients was balanced.
  Participants | 23 | 29 | 52
Ave PSA before radiotherapy [Median (Inter-Quartile Range); unit: ng/mL] | 0.34 [0.19 to 1.08] | 0.34 [0.13 to 0.95] | 0.34 [0.17 to 1.05]

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival
Description: Definition of failure is: serum PSA value of 0.2ng/mL or more above the postradiotherapy nadir followed by another higher value, a continued rise in the serum PSA despite radiotherapy (RT), initiation of systemic therapy after completion of RT, or clinical progression.
Time Frame: 3-Year post-intervention
Population: This outcome evaluated the failure-free survival difference (among those who received radiotherapy) between the trial group (in which FACBC PET scan was used) versus the control group (in which conventional-only imaging was used).
  FACBC PET Group: 83 enrolled subjects minus 3 withdrawals minus 4 patients not receiving radiotherapy due to PET findings = 76 participants.
  Conventional Imaging Group: 82 enrolled minus 1 withdrawal = 81 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
Percentage of participants | 75.5 | 63.0

2. Secondary Outcome: Decision Changes Regarding Radiotherapy Versus no Radiotherapy
Description: Number of decision changes regarding radiotherapy versus no radiotherapy based on F-Fluciclovine PET/CT guidance. This outcome was assessed immediately after the consensus reading of the Fluciclovine PET/CT was completed by nuclear medicine, an average of 1 week post intervention.
Time Frame: Average of 1 week post-intervention
Population: This outcome evaluated number of decision changes regarding the overall use of radiotherapy in the FACBC PET scan group only.
Measure: Number; unit: Number of decision changes
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 83 | 0
Number of decision changes | 4 |

3. Secondary Outcome: Decision Changes Regarding Whole-pelvis Versus Local Fields
Description: Number of decision changes regarding whole-pelvis versus local fields. This outcome was assessed immediately after the consensus reading of the Fluciclovine PET/CT was completed by nuclear medicine, an average of 1 week post intervention.
Time Frame: Average of 1 week post-intervention
Population: This outcome evaluated number of decision changes regarding changes from whole-pelvis to local fields and vice versa (local fields to whole pelvis) in the FACBC PET scan group only.
Measure: Number; unit: Number of decision changes
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 83 | 0
Number of decision changes | 24 |

4. Secondary Outcome: Total Number of Decision Changes
Description: Total number of radiotherapy decision changes regarding radiotherapy vs no radiotherapy and regarding whole pelvis vs local fields. This outcome was assessed immediately after the consensus reading of the Fluciclovine PET/CT was completed by nuclear medicine, an average of 1 week post intervention.
Time Frame: Average of 1 week post-intervention
Population: This outcome evaluated number of all radiotherapy-related decision changes in the FACBC PET scan group only.
Measure: Number; unit: Number of decision changes
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 83 | 0
Number of decision changes | 28 |

5. Secondary Outcome: Prostate Bed Clinical Target Volume (CTV)
Description: Absolute volume pre- vs post-PET. This outcome was assessed after radiotherapy treatment planning was completed by radiation oncology, an average of 1 month post-intervention.
Time Frame: Average of 1 month post-intervention
Population: Note that no participants were analyzed in the Conventional group Post-PET since they did not receive the PET intervention.
  FACBC PET Group: 83 enrolled subjects minus 3 withdrawals minus 4 patients not receiving radiotherapy due to PET findings = 76 participants.
  Conventional Imaging Group: 82 enrolled minus 1 withdrawal = 81 participants.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
mL
  Pre-PET | 134.14 (45.60) | 137.18 (51.36)
  Post-PET: number analyzed (Participants) | 76 | 0
  Post-PET | 135.61 (45.51) |

6. Secondary Outcome: Prostate Bed Planning Target Volume (PTV)
Description: Absolute volume were measured pre- vs post-PET. This outcome was assessed after radiotherapy treatment planning was completed by radiation oncology, an average of 1 month post-intervention.
Time Frame: Average of 1 month post-intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
mL
  Pre-PET | 324.50 (79.82) | 327.71 (88.61)
  Post-PET: number analyzed (Participants) | 76 | 0
  Post-PET | 329.54 (81.34) |

7. Secondary Outcome: PTV Dosimetric Endpoints
Description: Standard radiotherapy dosimetric endpoints used to evaluate target coverage. Planning target volume (PTV) at V100 and V110 refer to %volume of the structure receiving 100% and 110% of the prescription dose, respectively, pre and post positron emission tomography (PET). This outcome was assessed after radiotherapy treatment planning was completed by radiation oncology, an average of 1 month post-intervention.
Time Frame: Average of 1 month post-intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of volume
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
percentage of volume
  PTV2/PTV, V100% pre PET | 96.98 (1.56) | 96.36 (1.67)
  PTV2/PTV, V100% post PET: number analyzed (Participants) | 76 | 0
  PTV2/PTV, V100% post PET | 96.62 (1.54) |
  PTV2/PTV, V110% pre PET | 2.60 (7.81) | 0.42 (1.89)
  PTV2/PTV, V110% post PET: number analyzed (Participants) | 76 | 0
  PTV2/PTV, V110% post PET | 1.09 (6.11) |

8. Secondary Outcome: Rectum Dosimetric Endpoints
Description: Standard radiotherapy dosimetric endpoints used to evaluate normal tissue doses, in this case, the rectum. V40 and V65 refer to the %volume of the structure receiving 40 Gy and 65 Gy, respectively, pre and post positron emission tomography (PET) volumes were compared. This outcome was assessed after radiotherapy treatment planning was completed by radiation oncology, an average of 1 month post-intervention.
Time Frame: Average of 1 month post-intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of volume
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
percentage of volume
  Rectum, V40 pre PET | 45.01 (10) | 45.03 (10.89)
  Rectum, V40 post PET: number analyzed (Participants) | 76 | 0
  Rectum, V40 post PET | 45.07 (9.78) |
  Rectum, V65 pre PET | 18.35 (7.78) | 19.31 (7.82)
  Rectum, V65 post PET: number analyzed (Participants) | 76 | 0
  Rectum, V65 post PET | 18.48 (7.78) |

9. Secondary Outcome: Bladder Dosimetric Endpoints
Description: Standard radiotherapy dosimetric endpoints are used to evaluate normal tissue doses, in this case, the bladder. V40 and V65 refer to the %volume of the structure receiving 40 Gy and 65 Gy, respectively, pre and post positron emission tomography (PET) volumes were compared. This outcome was assessed after radiotherapy treatment planning was completed by radiation oncology, an average of 1 month post-intervention.
Time Frame: Average of 1 month post-intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of volume
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
percentage of volume
  Bladder, V40 pre-PET | 68.92 (14.94) | 68.95 (18.04)
  Bladder, V40 post-PET: number analyzed (Participants) | 76 | 0
  Bladder, V40 post-PET | 69.10 (14.70) |
  Bladder, V65 pre-PET | 49.68 (17.31) | 50.99 (19.35)
  Bladder, V65 post-PET: number analyzed (Participants) | 76 | 0
  Bladder, V65 post-PET | 50.29 (19.92) |

10. Secondary Outcome: Rate of ≥ Grade 2 GU (Genitourinary [Renal or Urinary]) Toxicity
Description: Provider-reported maximum acute (<90 days Post-Intervention) and late (≥90 days and up to 3-Years post-intervention) genitourinary toxicity based on CTCAE v4.0 criteria.
Time Frame: 3-Year post-intervention
Population: All patients in both the FACBC PET scan and the Conventional-imaging only groups.
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 83 | 82
Participants
  Number of patients with Acute GU toxicity | 18 | 21
  Number of patients with Late GU toxicity | 36 | 42

11. Secondary Outcome: Rate of ≥ Grade 2 GI (Gastrointestinal) Toxicity
Description: Provider-reported maximum acute (<90 days Post-Intervention) and late (≥90 days and up to 3-Years post-intervention) gastrointestinal toxicity ≥ Grade 2 based on CTCAE v4.0 criteria.
Time Frame: 3-Year post-intervention
Population: All patients in both the FACBC PET scan and the Conventional-imaging only groups.
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 83 | 82
Participants
  Number of patients with Acute GI toxicity | 16 | 11
  Number of patients with Late GI toxicity | 6 | 10

12. Secondary Outcome: Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC) GU (Genitourinary) Domain Score
Description: Patient-reported maximum genitourinary toxicity based on standard EPIC-CP questionnaire. EPIC GU domain score has a total score range 0-12. Higher score correlates with worse outcome. EPIC GU score includes the incontinence domain score and the irritative/obstructive.
Time Frame: 3-Year post-intervention
Population: Radiotherapy-treated patients in both the FACBC PET scan and the Conventional-imaging only groups.
  FACBC PET Group: 83 enrolled subjects minus 3 withdrawals minus 4 patients not receiving radiotherapy due to PET findings = 76 participants.
  Conventional Imaging Group: 82 enrolled minus 1 withdrawal = 81 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
score on a scale
  EPIC GU-incontinence domain score | 2.99 (3.10) | 3.50 (3.02)
  EPIC GU - irritative/obstructive | 1.80 (2.02) | 2.66 (2.70)

13. Secondary Outcome: Expanded Prostate Cancer Index Composite (EPIC) GI (Gastrointestinal) Domain Score
Description: Patient-reported maximum gastrointestinal toxicity based on standard EPIC-CP questionnaire. Total score range 0-12. Higher score correlates with worse outcome.
Time Frame: 3-Year post-intervention
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
score on a scale | 1.20 (1.99) | 1.41 (2.21)

14. Secondary Outcome: Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain Score
Description: Patient-reported maximum sexual function toxicity based on standard EPIC-CP questionnaire. Total score range 0-12. Higher score correlates with worse outcome.
Time Frame: 3-Year post-intervention
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
score on a scale | 6.04 (4.14) | 7.37 (3.79)

15. Secondary Outcome: Expanded Prostate Cancer Index Composite (EPIC) Total Score
Description: Patient-reported maximum overall (genitourinary, gastrointestinal, and sexual function) toxicity based on standard EPIC-CP questionnaire. Total score range 0-60. Higher score correlates with worse outcome.
Time Frame: 3-Year post-intervention
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
Number analyzed (Participants) | 76 | 81
score on a scale | 13.90 (9.98) | 17.02 (9.78)

ADVERSE EVENTS:
Time Frame: Up to 3-years post-intervention
Description: Severe Adverse Events (SAEs) were defined as any provider-reported grade 3 or higher Gastrointestinal [GI] or Genitourinary [GU] toxicity. Acute toxicity was measured <90 days Post-Intervention and late toxicity was measured ≥90 days and up to 3-Years post-intervention.
  Adverse Events (AE's) were defined as any provider-reported (acute or late) grade 2 toxicity.
Arm/Group | FACBC PET Scan | Conventional-Only Imaging
All-Cause Mortality (participants affected / at risk) | 1/83 | 1/82
Serious Adverse Events (participants affected / at risk) | 5/83 | 8/82
Other Adverse Events (participants affected / at risk) | 71/83 | 76/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FACBC PET Scan (N=83) | Conventional-Only Imaging (N=82)
Hematuria - Acute (Renal and urinary disorders) | 0 (0) | 3 (3)
Hematuria - Late (Renal and urinary disorders) | 5 (5) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FACBC PET Scan (N=83) | Conventional-Only Imaging (N=82)
Diarrhea (Gastrointestinal disorders) | 22 (22) | 21 (21)
Urinary Frequency (Renal and urinary disorders) | 49 (49) | 55 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT01666808/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT01666808/ICF_002.pdf